CLINICAL TRIAL: NCT04921254
Title: A Phase 1, Double-blinded, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of BSG005 Following Single and Multiple Ascending Doses in Healthy Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of BSG005.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biosergen AS (Industry)
Collaborators: Select Pharma Pty Ltd (Unknown); Greenlight Clinical (Unknown); Nucleus Network Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSG1.01
Record Dates: First submitted 2021-04-24; First posted 2021-06-10 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Invasive Fungal Infections
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Intervention Model Description: Single escalation dose safety, tolerability and PK followed by multiple escalation dose for safety, tolerability and PK.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: DB and placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BSG005 (Experimental): Active antifungal drug
  Interventions: Drug: BSG005 or placebo
- Placebo (Placebo Comparator): Will be a 5% glucose infusion
  Interventions: Drug: BSG005 or placebo

INTERVENTIONS:
Drug: BSG005 or placebo — SAD part is a single IV infusion of ascending doses of BSG005 or placebo - a 30 minutes infusion that may be extended to 2 hours if infusion reactions occur.
  The MAD part is single daily infusions of the cohort dose over 30 minutes (that may be delayed up to 2 hours in case of infusion reactions) and which will be repeated daily for 7 days. Objective is safety, tolerability and PK on day 1 and day 7 and to establish steady state plasma level.
  Other Names: BSG005; Placebo

SUMMARY:
A Phase 1, double-blinded, placebo-controlled study to assess the safety, tolerability, and pharmacokinetics of BSG005 following single and multiple ascending doses in healthy subjects. The study will include a single ascending dose part and a multiple ascending dose part

DETAILED DESCRIPTION:
The study will investigate the safety and tolerability of BSG005 in healthy subjects. The study will also include pharmacokinetic investigations.

There will be an ascending single dose part (SAD) with 6 subject in a study dose cohort of which 2 will be placebo and 4 will be on active drug. This concept will be replicated in the multiple ascending dose (MAD) part.

There is expected to be up to6 cohorts in SAD part with a starting dose calculated from the GLP NOAEL dose levels and from that increasing dose levels will be tested after a Safety Review Committee (SRC) has approved the escalation to next dose level. The key parameters are infusion reactions, kidney, liver and potassium changes during and after administration of BSG005.

Depending on the outcome of the SAD part the MAD part may include 4 or 5 dose levels administered daily over 7 days. Key parameters are the same as in the SAD part but extended to cover monitoring over 14 days. Pharmacokinetics at day 1 and day 7 will be investigated.

Key evaluation is on safety and tolerability during and after 7 days of dosing and pharmacokinetic investigations and the steady state plasma levels.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, each individual must satisfy all the following criteria:

1. Male adult subjects aged 18 - 55 years at screening.
2. Subjects without concurrent illnesses who do not require any medical treatments.
3. Judged by an Investigator to be in good health as documented by the medical history, physical examination (including but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory, and central nervous systems), 12-lead ECG, vital sign assessments, clinical laboratory assessments, and by general observations. Any abnormalities or deviations outside the normal ranges for any of clinical testing (laboratory tests, ECG, vital signs) can be repeated at the discretion of the Investigator(s) and/or judged to be not clinically significant for study participation.
4. Body Mass Index ≥18 and <30 kg/m2 and a weight of at least 50 kg.
5. Negative drug and alcohol screen in urine. Negative pregnancy test (females)
6. Subject is a non-smoker or smokes ≤ 10 cigarettes per day (or equivalent).
7. Must be able and willing to provide written informed consent.
8. Are willing to remain in the study unit for the entire duration of the treatment period, attend all scheduled visits, and comply with all study procedures.
9. If sexually active males, must use a condom OR abstinence OR same sex partner OR surgically sterile OR partner is of non-childbearing potential.

Exclusion Criteria:

If an individual meets any of the following criteria, he or she is ineligible for this study:

1. Participation in any study involving an investigational drug or device within the past 30 days or ongoing participation in a study with an investigational drug or device.
2. Any clinical evidence that the Investigator feels would place the subject at increased risk with the investigational product.
3. Subject shows clinically significant abnormalities in physical examination, vital signs, 12-lead ECG, or clinical laboratory parameters for the screening assessments (especially for liver enzymes, and serum creatinine and estimated creatinine clearance) according to the Investigator's judgment.
4. Has liver enzyme results (AST, ALT, GGT) above the upper normal limit (UNL): AST 37 U/L; ALT 78 U/L; GGT 55 U/L.
5. Has a creatinine value outside the normal range (female <0.51 mg/dL; male <0.67 mg/dL) and an estimated creatinine clearance (Cockcroft-Gault) < 30 mL/min
6. Subject with, or history of clinically significant neurologic, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, or other major disorders.
7. Subject who has a sitting or lying blood pressure at screening, after resting for at least 5 minutes: systolic blood pressure > 155 or < 90 mmHg, or diastolic blood pressure > 90 or < 40 mmHg.
8. Subject who has a sitting or lying pulse rate at screening, after resting for at least 5 minutes, outside the range of < 39 or > 101 beats/min.
9. Subject who donated blood or who had a comparable blood loss (approximately 500 mL) during the last 30 days prior to start of this study.
10. Subject with a known history of clinically significant drug allergies in the opinion of the Investigator or with a known allergy to any medicine chemically related to the study medication.
11. Subject who has had a clinically significant illness within four weeks prior to screening in the opinion of the Investigator.
12. Subject with a history of chronic alcohol (regular daily intake of more than, e.g., three standard drinks) or drug abuse within the last 6 months prior to first administration or evidence of such abuse as indicated by the laboratory profile conducted during the screening examination.
13. Subject who has received prescription drugs or OTC medication other than dietary supplements, occasional ibuprofen, standard dose vitamins, or herbal products within 2 weeks prior to the first administration (with the exception of up to 1000 mg acetaminophen per day).
14. Subject who plans to take concomitant medications while enrolled in the study (with the exception of up to 1000 mg acetaminophen per day or vitamins, dietary supplements, or herbal products).
15. Subject who received any treatment agents known to alter the major organs or systems within 30 days prior to the first administration (e.g., diuretics, nephro- or liver toxic medication, barbiturates, phenothiazines, cimetidine, more than 1.0 L of caffeine-containing beverages per day, etc.).
16. Subject who has consumed any grapefruit containing product on the day of clinic check-in.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only males as repro tox is only ongoing.
Enrollment: 72 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
AE recorded during and after BSG005 infusion | On single dose(-1 to 7 days) and multiple dosing (- 1 to 14 days) changes.
  The Investigator will carefully monitor each subject throughout the study for any AEs (coded to preferred term and system organ class using the Medical Dictionary for Regulatory Activities [MedDRA])

SECONDARY OUTCOMES:
Pharmacokinetics of BSG005 infusion at different dose levels in SAD and MAD conditions | 24 hours.
  Area under the concentration-time curve from time 0 (predose) to time 24 hours.
Cmax | 24 hours
  Maximum concentration (Cmax)
Tmax | 24 hours
  Time to reach maximum concentration (Tmax)
AUC (0-t) | 24 hours
  Area under concentration-time curve from time 0 (predose) to the last quantifiable data point (AUC(0-t))
t1/2 | 24 hours
  Terminal half-life (t1/2)
Steady state concentration | 8 days
  concentration on day 7 at pre-dose and at 24 hours on day 8 in MAS part

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Ryan, MD, Principal Investigator — Nucleus Network, Melbourne site, Australia
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No